CLINICAL TRIAL: NCT00244621
Title: A Dose-ranging Safety and Pharmacokinetics Study of Candesartan Cilexetil in Hypertensive Pediatric Subjects 1 to Less That 6 Years of Age: A 4-week, Multicenter, Randomized, Double-blind Study With a 1-year, Open-label, Follow-up Period.
Brief Title: Atacand Dose Ranging in Hypertensive Pediatric Subjects 1 Year to Less Than 6 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2451C00002; 328
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2009-09-15 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Hypertension
Keywords: Pediatric hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Experimental): 0.05 mg/kg Atacand oral liquid dose
  Interventions: Drug: candesartan cilexetil (Atacand)
- 2 (Experimental): 0.20 mg /kg Atacand oral liquid dose
  Interventions: Drug: candesartan cilexetil (Atacand)
- 3 (Experimental): 0.40 mg /kg Atacand oral liquid dose
  Interventions: Drug: candesartan cilexetil (Atacand)

INTERVENTIONS:
Drug: candesartan cilexetil (Atacand) — 0.05 mg/kg once daily oral liquid dose
  Other Names: Atacand
  Arms: 1
Drug: candesartan cilexetil (Atacand) — 0.20 mg/kg once daily oral liquid dose
  Other Names: ATACAND
  Arms: 2
Drug: candesartan cilexetil (Atacand) — 0.40 mg/kg once daily oral liquid dose
  Other Names: ATACAND
  Arms: 3

SUMMARY:
This is a dose ranging study of candesartan cilexetil in hypertensive pediatric subjects ages 1 to less than 6 years of age. It employs a double blind, randomized, dose ranging design intended for conduct as a multicenter trial. There are 3 study 'periods': a 1-week placebo run-in, a 4-week double blind treatment, and a 52-week open-label, long-term treatment period. Subjects undergo a screening evaluation, then a 1-week single-blind, placebo run-in, after which eligible subjects are allocated to receive 1 of 3 dose levels of candesartan cilexetil (0.05 mg/kg, or 0.20 mg /kg or 0.40 mg /kg), liquid formulation, in a 1:1:1 ratio for 4-weeks. At the end of randomized dose allocation (Day 28), blood pressure assessment will be performed and subjects may begin the 52-week, open-label treatment period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by a parent or a legal guardian.
* Weight > 10 kg and < 40 kg.
* SiSBP and/or SiDBP > 95th percentile and < 20 mm Hg (systolic) and/or 10 mm Hg (diastolic) above the 95th percentile at screening and at randomization based on height-adjusted charts for age and gender.

Exclusion Criteria:

* Any situation, clinical condition or laboratory abnormality that, in the opinion of the investigator or sponsor, may interfere with the subject's participation in the study or would pose a significant risk to the subject or interfere with the assessment of safety and efficacy endpoints.
* Weight < 10 kg and > 40 kg.
* Less than 80% compliance with study medication during single-blind placebo screening as assessed by residual medication volume.
* Hypertension secondary to pheochromocytoma, hyperthyroidism, or Cushing's Syndrome.
* Uncorrected coarctation of the aorta, bilateral renal artery renal artery stenosis in a single kidney.
* Estimated glomerular filtration rate (GFR) < 50 mL/min/1.73m 2 based on the Schwartz Formula (Schwartz et al, 1987).
* Renal transplant < 6 months prior to study entry. Subjects who have received a renal transplant > 6 months prior to study entry may participate in the study if: 1) renal function is stable, 2) estimated GFR >50 mL/min/1.73m 2, 3) stable doses of immunosuppressive medications are anticipated throughout the 4-week, double-blind period of the study, 4) no episodes of acute allograft rejection have occurred within 30 days of study entry, and 5) the renal allograft has no documented renal artery stenosis.

Nephrotic syndrome not in remission.

* Unstable insulin dependent diabetes mellitus.
* Known bleeding, coagulation, or platelet disorder that could interfere with blood sampling.
* Clinically significant valvular heart disease.
* Clinical diagnosis of heart failure.
* Clinically significant arrhythmia (eg, any arrhythmia requiring medical therapy or that causes symptoms).
* Second or third degree AV block.
* Impaired liver function defined as either acute liver disease or chronic liver disease with persistent liver enzyme values greater than 1½ times the upper limit of the reference range for aspartate aminotransferase (AST) or alanine aminotransferase (ALT).
* Known hypersensitivity to ARBs.
* Currently receiving an angiotensin receptor blocker or an angiotensin converting enzyme inhibitor that in the investigator's judgment cannot safely be withdrawn during the study.
* Subjects receiving an angiotensin receptor blocker or an angiotensin converting enzyme inhibitor may be eligible if they undergo withdrawal of the antihypertensive medication over a 2-week washout period and subsequently meet BP inclusion/exclusion criteria.
* Subjects currently receiving other classes of antihypertensive medications (eg, diuretics, calcium channel blockers or beta-blockers) and whose BP values meet inclusion/exclusion criteria may participate in the study while continuing their current antihypertensive medication regimen. Up to 2 concomitant antihypertensive medications are permitted. Doses and dose regimens of concomitant antihypertensive medications must remain unchanged during the 4-week double-blind period of the study.
* Currently using, or used within 14 days prior to receiving double-blind medication, any concomitant medications which in the opinion of the investigator could negatively affect the subject.
* Unable or unwilling to comply with the study requirements including blood sampling and swallowing study drug suspension.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2004-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Atacand Medical Science Director, MD, Study Director — AstraZeneca
Locations (38):
- United States (16):
  - Research Site, Birmingham, Alabama
  - Research Site, Little Rock, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Boise, Idaho
  - Research Site, Detroit, Michigan
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Malvern, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Beaumont, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
- Belgium (2):
  - Research Site, Edegem
  - Research Site, Ghent
- Research Site, Aarhus, Denmark
- Research Site, Strasbourg, France
- Germany (6):
  - Research Site, Berlin
  - Research Site, Erlangen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Marburg
  - Research Site, Rostock
- Italy (4):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Warsaw
- Research Site, San Juan, Puerto Rico
- Ukraine (2):
  - Research Site, Crimea
  - Research Site, Kyiv
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

REFERENCES:
- [Derived] Schaefer F, van de Walle J, Zurowska A, Gimpel C, van Hoeck K, Drozdz D, Montini G, Bagdasorova IV, Sorof J, Sugg J, Teng R, Hainer JW; Candesartan in Children with Hypertension Investigators. Efficacy, safety and pharmacokinetics of candesartan cilexetil in hypertensive children from 1 to less than 6 years of age. J Hypertens. 2010 May;28(5):1083-90. doi: 10.1097/HJH.0b013e328336b86b. PMID 20160654

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included male and female participants 1 to <6 years of age with mild to moderate hypertension. The participants were recruited during the time period from 04 November 2004 to 07 August 2008 at pediatric clinics in the USA, Puerto Rico and Europe.
Pre-assignment Details: One to 2 weeks following a screening evaluation, participants underwent a 1-week, single-blind, placebo run-in period to reduce the variability in the baseline blood pressure measurements and to stabilize any concurrent antihypertensive medications.
Groups:
- Atacand .05 mg: candesartan cilexetil (Atacand) 0.05 mg/kg once daily oral liquid dose
- Atacand .20 mg: candesartan cilexetil (Atacand) 0.20 mg/kg once daily oral liquid dose
- Atacand .40 mg: candesartan cilexetil (Atacand) 0.40 mg/kg once daily oral liquid dose
Period: Double-blind Treatment Period
Arm/Group | Atacand .05 mg | Atacand .20 mg | Atacand .40 mg
Started | 29 | 32 | 32
Completed | 27 | 29 | 30
Not Completed | 2 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Multiple Reasons | 2 | 1 | 1
Period: Open-label Treatment Period
Arm/Group | Atacand .05 mg | Atacand .20 mg | Atacand .40 mg
Started | 26 (One participant discontinued study due to Adverse Event after completing the double-blind period.) | 29 | 30
Completed | 25 | 28 | 28
Not Completed | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Moved abroad | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atacand .05 mg | Atacand .20 mg | Atacand .40 mg | Total
Number analyzed (Participants) | 29 | 32 | 32 | 93
Age, Customized [Number; unit: Participants]
  1 to <2 years | 6 | 5 | 5 | 16
  2 to <6 years | 23 | 27 | 27 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 12 | 33
  Male | 18 | 22 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 4 in Systolic Blood Pressure (SBP)
Time Frame: From randomisation to end of double-blind treatment (4 weeks)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Atacand .05 mg | Atacand .20 mg | Atacand .40 mg
Number analyzed (Participants) | 29 | 32 | 32
mm Hg | -6.0 (9.4) | -8.9 (9.2) | -12.0 (8.3)

2. Secondary Outcome: Mean Change From Baseline to Week 4 in Diastolic Blood Pressure (DBP)
Time Frame: From randomisation to end of double-blind treatment (4 weeks)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Atacand .05 mg | Atacand .20 mg | Atacand .40 mg
Number analyzed (Participants) | 29 | 32 | 32
mm Hg | -5.2 (6.7) | -7.9 (12.9) | -11.1 (9.2)

3. Secondary Outcome: Change in Albumin/Creatinine (A/C) Ratio for Each Assigned Dose Level From Baseline to Day 28
Time Frame: From randomisation to day 28
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Atacand .05 mg | Atacand .20 mg | Atacand .40 mg
Number analyzed (Participants) | 19 | 19 | 19
Percent change | -11.1 [-42.5 to 33.3] | -40.6 [-68.1 to 25.0] | -50.0 [-68.9 to 15.8]

4. Secondary Outcome: Change in Protein/Creatinine (P/C) Ratio for Each Assigned Dose Level From Baseline to Day 28
Time Frame: From randomisation to day 28
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Atacand .05 mg | Atacand .20 mg | Atacand .40 mg
Number analyzed (Participants) | 25 | 26 | 27
Percent change | 0.0 [-25.0 to 50.0] | -29.2 [-50.0 to 0.0] | 0.0 [-40.7 to 0.0]

ADVERSE EVENTS:
Arm/Group | Atacand .05 mg | Atacand .20 mg | Atacand .40 mg
Serious Adverse Events (participants affected / at risk) | 6 | 5 | 4
Other Adverse Events (participants affected / at risk) | 0/29 | 0/32 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Atacand .05 mg | Atacand .20 mg | Atacand .40 mg
Lymphadenitis (Blood and lymphatic system disorders) | 0/29 | 1/32 | 0/32
Catheter Site Haematoma (Blood and lymphatic system disorders) | 1/29 | 0/32 | 0/32
Catheter Site Necrosis (Blood and lymphatic system disorders) | 1/29 | 0/32 | 0/32
Pyrexia (Blood and lymphatic system disorders) | 0/29 | 1/32 | 1/32
Drug Hypersensitivity (Immune system disorders) | 0/29 | 0/32 | 1/32
Bronchiolitis (Infections and infestations) | 1/29 | 0/32 | 0/32
External Ear Cellulitis (Infections and infestations) | 1/29 | 0/32 | 0/32
Pneumonia (Infections and infestations) | 1/29 | 0/32 | 0/32
Pneumonia Parainfluenzae Viral (Infections and infestations) | 0/29 | 1/32 | 0/32
Pyelonephritis (Infections and infestations) | 1/29 | 0/32 | 0/32
Upper Respiratory Tract Infection (Infections and infestations) | 0/29 | 1/32 | 0/32
Urinary Tract Infection (Infections and infestations) | 0/29 | 2/32 | 2/32
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0/29 | 1/32 | 0/32
Glomerulonephritis Chronic (Renal and urinary disorders) | 0/29 | 0/32 | 1/32
Nephrotic Syndrome (Renal and urinary disorders) | 1/29 | 0/32 | 0/32
Vena Cava Thrombosis (Vascular disorders) | 1/29 | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days